CLINICAL TRIAL: NCT02777216
Title: ConfidenHTTM System Safety and Performance of Diagnostic Electrical Mapping of Renal Nerves in Hypertensive Patients and/or Potential Candidates for a Renal Sympathetic Denervation (RDN) Procedure
Brief Title: ConfidenHT System for Diagnostic Electrical Mapping of Renal Nerves
Acronym: RDN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: BlueWind Medical (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 167CLP
Record Dates: First submitted 2016-05-17; First posted 2016-05-19 (Estimated); Last update posted 2018-02-26 (Actual); Status verified 2017-12

CONDITIONS: Hypertension
Keywords: RDN
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- ConfidenHT system (Experimental): ConfidenHT system
  Interventions: Device: ConfidenHT system

INTERVENTIONS:
Device: ConfidenHT system — ConfidenHT Medical system
  Other Names: ConfidenHT Medical system

SUMMARY:
To evaluate the safety and performance of the ConfidenHT System

DETAILED DESCRIPTION:
To evaluate the safety and performance of the ConfidenHT System for diagnostic mapping of renal nerves; functional distribution of renal nerves and the effect of renal nerve stimulation on the blood pressure

ELIGIBILITY:
Inclusion Criteria:

1. Signed written informed consent.
2. Age >18 years and <75.
3. Either:

   1. Hypertensive patients planned to undergo elective cardiac catheterization
   2. Potential candidates for renal sympathetic denervation
4. Main renal artery with diameter ≥ 4.0mm.
5. Glomerular Filtration Rate (GFR) >45 mL/min
6. A patient who is mentally competent with the ability to understand and comply with the requirements of the study.
7. The patient agrees to attend all follow-up evaluations and is willing to complete required exams and tests.
8. Female patients with childbearing potential must agree:

   * to use a valid method of contraception (oral contraceptives, intrauterine device, subcutaneous contraceptive implant, vaginal ring)
   * to perform a pregnancy test

Exclusion criteria:

1. Previous participation in another study with any investigational drug or device within the past 30 days.
2. Relevant renal artery disease (% diameter stenosis>30%, aneurysm or fibromuscular dysplasia).
3. Known secondary causes of hypertension.
4. The patient has a life expectancy ≤ 12 months.
5. The patient has undergone prior renal denervation, renal stenting, and/or abdominal aortic stent grafts.
6. The patient has chronic oxygen use other than nocturnal support for sleep apnea.
7. The patient has type I diabetes mellitus.
8. The patient has had a previous organ transplant or is awaiting a renal transplant.
9. Active implantable medical device (e.g. ICD or CRT-D; neuromodulator/spinal stimulator; baroreflex stimulator).
10. The patient has triple ipsilateral artery ostia.
11. Moderate to severe valvular heart disease.
12. The patient has other concomitant conditions that may adversely affect the patient or the study outcome.
13. Female who is pregnant, nursing or planning to become pregnant.
14. Documented contraindication or allergy to contrast medium not amenable to treatment.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2016-10 (Actual); Primary Completion 2017-11 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
The incidence of serious adverse events (system and/or procedure related events) | 3 months
  The incidence of serious adverse events (system and/or procedure related events)

CONTACTS AND LOCATIONS:
Overall Officials: Kostas Tsioufis, MD, Principal Investigator — Hippocratio Hospital, Athens, Greece
Locations (3):
- Hippocratio Hospital, Athens, Greece
- Netherlands (2):
  - EMC, Rotterdam
  - UMC, Utrecht

IPD SHARING:
Plan to Share IPD: No